CLINICAL TRIAL: NCT03241992
Title: Utility of MyChart for Improving Quality of Life and Patient Satisfaction in Patients With Inflammatory Bowel Disease.
Brief Title: MyChart in Patients With Inflammatory Bowel Disease.
Acronym: MyIBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Jason Reich, Fellow, Gastroenterology. General Internal Medicine Department, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-35695
Record Dates: First submitted 2017-08-04; First posted 2017-08-08 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Inflammatory Bowel Disease; IBD; Electronic Health Record; Patient Portal; Quality of Life
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MyChart Intervention (Experimental): Subjects in the control arm will be enrolled in MyChart during the consent process and receive MyChart Disease Specific targeted IBD information and reminders as well as mood questionnaires. At week 2 subjects will receive reminders to get vaccinated with another reminder sent at 3 months. At month 1, subjects will receive the Promis Adult Short Form questionnaires for depression and anxiety through MyChart. If a subject is identified as having mild, moderate or a severe mood disorder a message will be sent to their gastroenterologist with a recommendation to discuss the results with the patient and to consider a referral to mental health services. Subjects will also receive educational information about IBD every 6 weeks along with reminders to take their medications.
  Interventions: Behavioral: MyChart Disease Specific
- Usual Care (No Intervention): Subjects in the control arm will be enrolled in MyChart during the consent process if they are not previously enrolled. Enrollment in MyChart will provide them with access to their medical record and the ability to send or receive messages with their gastroenterologist or any other providers they see at our institution. For patients with IBD it is standard practice to discuss medication adherence, vaccinations, and their mood at each appointment. Subjects will receive generic, non-IBD related messages through MyChart.

INTERVENTIONS:
Behavioral: MyChart Disease Specific — Subjects receive targeted IBD information and reminders as well as mood questionnaires.
  Arms: MyChart Intervention

SUMMARY:
This study will be the first to assess the use of an electronic health records patient portal for patients with Inflammatory Bowel Disease. Patients with Inflammatory Bowel Disease (IBD), have reduced quality of life, high rates of depression and anxiety, do not receive routine preventative health maintenance (such as vaccines) at the same rate as the general public, and have low adherence to medications. The investigators are seeking to understand whether an electronic health record patient portal (EPIC's MyChart), can be utilized to improve quality of life in this patient population.

DETAILED DESCRIPTION:
This study will be a single site randomized control trial.

Patients will be randomized into a control arm and intervention arm. At baseline the investigators will obtain demographic data, quality of life measures, and satisfaction with MyChart for those patients who are alrealy active portal users. The control arm will receive periodic messages through MyChart that are not specific to IBD. The intervention arm will receive more specific disease related information such as IBD educational information, reminders to take their medications, and reminders to get vaccinated. The intervention arm will also receive questionnaires that assess their mood (depression and anxiety). The investigators will then inform the primary gastroenterologist for those patients in whom mild, moderate or severe depression and anxiety is identified. At the end the study, in both groups investigators will measure quality of life as measured by the Short Inflammatory Bowel Disease Questionnaire (SIBDQ), a validated questionnaire for measuring health-related quality of life in patients with Crohn's and Ulcerative Colitis. Secondary outcomes will include: Satisfaction with Mychart as measured by a MyChart satisfaction survey, time to referral to mental health provider for patients identified with mild, moderate, or severe depression, or anxiety (PROMIS Depression and Anxiety Questionnaires), and Vaccine uptake (using a simple yes/no questionnaire asking patients if they received Flu, PCV13 or PPSV23.

The findings of this study will allow future clinicians to better understand how a patient portal can be utilized as a tool for the management of patients with IBD. This findings may lead to increased physician and patient engagement with the MyChart patient portal.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women 18 years and older with a diagnosis of Inflammatory Bowel Disease (Crohn's or Ulcerative Colitis, or Indeterminate Colitis by standard criteria) who are scheduled for an upcoming appointment at the outpatient gastroenterology clinic or infusion unit.

Exclusion Criteria:

* Non-English speaking patients
* Patients identified by their physicians as being too cognitively impaired to participate
* Patients without access to computer with internet
* Patients not expected to be in the study area for the duration of the study such as patients only seen for a one time second opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-01-20 (Actual)

PRIMARY OUTCOMES:
Quality of life based on the SIBDQ | 6 months
  Quality of life will be measured using the Short Inflammatory Bowel Disease Questionnaire (SIBDQ) which is a 10 item health-related quality of life (HRQoL) tool measuring physical, social, and emotional status (scores can range from 10-70, poor to good HRQoL).

SECONDARY OUTCOMES:
Satisfaction with MyChart | 6-months
  The 14 item embedded MyChart Satisfaction Survey will be used to measure satisfaction. Responses for 12 of the questions are answered on a scale of 0 to 10 where 10=Strongly Agree, 5=Neither Agree nor Disagree, and 0=Strongly Disagree, so the higher the score for those questions the greater the satisfaction. there is also a question about the number of times myChart was used and an open-ended comments question..
Influenza vaccine uptake | 6-months
  To measure vaccine uptake for flu the patients will be asked if they received the flu shot in the previous year. A chart review will be done to confirm the self reported information.
Pneumococcal pneumonia (PCV13, PPSV23) vaccine uptake | 6-months
  To measure PCV13, PPSV23 vaccine uptake for pneumococcal pneumonia the patients will be asked if they received the vaccine in the previous year. A chart review will be done to confirm the self reported information.
Time to Referral for Behavioral Health | 6-months
  After a patient has been identified as having anxiety or depression and a message has been sent to their healthcare provider the time it takes the provider to refer the patient to behavioral health will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Reich, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No